CLINICAL TRIAL: NCT01898000
Title: "Triphala" - A New Herbal Mouthwash in Gingivitis: A Randomized Controlled Clinical Trial
Brief Title: "Triphala" - A New Herbal Mouthwash in Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2011-2012
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Gingivitis
Keywords: Gingivitis; Herbal medicine; Plaque control
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Behavioral: Triphala mouthwash — Subjects were instructed to use 15ml mouthwash twice daily and were instructed not to rinse/eat anything for 30 min after mouthwash use. Subjects were also asked to refrain from all other unassigned forms of oral hygiene aids, including dental floss and chewing gum during the study. No oral hygiene instructions like brushing and flossing were given to the subjects to exclude the influence of improved oral hygiene practices on the results.
Behavioral: Chlorhexidine mouthwash — Subjects were instructed to use 15ml mouthwash twice daily and were instructed not to rinse/eat anything for 30 min after mouthwash use. Subjects were also asked to refrain from all other unassigned forms of oral hygiene aids, including dental floss and chewing gum during the study. No oral hygiene instructions like brushing and flossing were given to the subjects to exclude the influence of improved oral hygiene practices on the results.

SUMMARY:
The present study was a randomized control clinical trial, which included 90 subjects with chronic generalised gingivitis of age group 25-40 years, reporting to outpatient department of Periodontics, Government Dental College & Research Institute, Bangalore form January 2013 to April 2013. The research protocol was initially submitted and approved by the Institutional Ethical Committee and Review Board of the Government Dental College and Research Institute, Bangalore. After ethical approval, all subjects were verbally informed and written signed informed consent was taken for participation in the study.

Ninety subjects diagnosed with chronic generalized gingivitis were randomly assigned into three groups: Group I: Placebo mouthwash, Group II: Triphala (TRP) mouthwash, Group III: Chlorhexidine (CHX) mouthwash. Subjects were instructed to use mouth wash twice daily. The plaque index (PI), gingival index (GI) and oral hygiene index- simplified (OHI-S) and microbiological colony counts were recorded on baseline (B/L) and 7, 30 and 60 days respectively.

TRP mouthwash was found to decrease the inflammatory parameters. As improvement in gingivitis was comparable to that of CHX mouthwash thus TRP mouthwash can be considered as a potential therapeutic agent in treatment of gingivitis.

DETAILED DESCRIPTION:
Objective: The aim of the present study is to evaluate the efficacy of triphala (TRP) as a mouthwash in reduction of plaque and gingivitis.

Material & Methods: Ninety subjects diagnosed with chronic generalized gingivitis were randomly assigned into three groups: Group I: Placebo mouthwash, Group II: TRP mouthwash, Group III: Chlorhexidine (CHX) mouthwash. Subjects were instructed to use mouth wash twice daily. The plaque index (PI), gingival index (GI) and oral hygiene index- simplified (OHI-S) and microbiological colony counts were recorded on baseline (B/L) and 7, 30 and 60 days respectively.

Results: There was a gradual decrease in the PI, GI and OHI-S scores by the 7 days, 30 days and 60 days time interval, respectively, in all three groups. Microbial counts also showed significant reduction in all the groups at all the time intervals except in Group 1. There was a significant difference with respect to reduction in PI, GI, OHI-S and microbiological counts in Group I as compared to Group II and Group III. However, no significant difference was found between Group II and Group III for all the parameters at all-time intervals.

Conclusion: TRP mouthwash was found to decrease the inflammatory parameters. As improvement in gingivitis was comparable to that of CHX mouthwash thus TRP mouthwash can be considered as a potential therapeutic agent in treatment of gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy subjects of 25-40 years of age with previously untreated gingivitis and minimum 20 teeth,
* gingival index > 1,
* pocket probing depth < 3 mm,
* clinical attachment loss = 0,
* with no evidence of radiographic bone loss

Exclusion Criteria:

* use of systemic antibiotics and anti-inflammatory drugs in the previous 6 months,
* known systemic disease,
* with orthodontic appliances or bridge work that would interfere with evaluation,
* allergy to ingredient used in the study,
* alcoholics,
* who use tobacco in any form,
* mentally retarded subjects,
* pregnant or
* lactating females and
* subjects with poor compliance

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Gingival Index (GI) | differences for the mean GI from B/L to 7 days, 30 and 60 days
  The primary outcome variable was the differences for the mean gingival Index (GI) from B/L to 7 days, 30 and 60 days.

SECONDARY OUTCOMES:
Change in Plaque Index (PI) | From Baseline (B/L) to 7 days, 30 and 60 days
  Differences in mean reduction in plaque index (PI) from baseline (B/L) to 7, 30 and 60 days

OTHER OUTCOMES:
Change in oral hygiene index simplified (OHI-S) | From baseline (B/L) to 7 days, 30 days and 60 days
  differences in mean reduction in Oral hygiene index simplified ( OHI-S)from baseline (B/L) to 7 days, 30 days and 60 days
Change in microbiological colony counts | From baseline (B/L) to 7 days, 30 days and 60 days
  in microbiological colony counts from baseline (B/L) to 7 days, 30 days and 60 days